CLINICAL TRIAL: NCT00705289
Title: Epidemiology, Correlation and Predictive Value of Disease Activity and Biomarkers in RA Patients Initiated on Infliximab in Clinical Practice
Brief Title: A Study to Observe Characteristics of Rheumatoid Arthritis in Patients Using Infliximab (Study P04250)
Acronym: REMARK
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04250
Record Dates: First submitted 2008-06-23; First posted 2008-06-26 (Estimated); Results first posted 2010-06-10 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and Urine samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- RA Subjects/ Infliximab 3 mg/kg: Subjects with rheumatoid arthritis (RA) in whom treatment with infliximab is started for the first time, in line with current clinical practice (and thus consistent with the European Summary of Product Characteristics [SPC] of Remicade®).
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab used in line with current clinical practice and local guidelines.
  Other Names: Remicade®; SCH 215596

SUMMARY:
This 14-week non-interventional study will observe patients with rheumatoid arthritis (RA) who are being treated with infliximab for the first time, in order to learn about their disease characteristics. Patients in this study will be treated for RA with infliximab and in a usual manner as decided by their physician.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with RA
* Physician has decided, with the subject's consent, to begin treatment with infliximab
* Written informed consent form signed by both the subject and the physician.

Exclusion Criteria:

* Subjects who have previously been exposed to infliximab

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be patients with rheumatoid arthritis in whom treatment with infliximab is started for the first time, in line with current clinical practice (and thus consistent with the European SPC of Remicade®).
  Subjects will be recruited from approximately 12 countries, including: Austria, Belgium, Denmark, France, Greece, the Netherlands, Norway, Poland, Portugal, Sweden, Switzerland and Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2005-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

REFERENCES:
- [Result] Westhovens R, van Vollenhoven RF, Boumpas DT, Brzosko M, Svensson K, Bjorneboe O, Meeuwisse CM, Srinivasan S, Gaudin P, Smolen JS, Rahman MU, Nelissen RL, Vastesaeger N. The early clinical course of infliximab treatment in rheumatoid arthritis: results from the REMARK observational study. Clin Exp Rheumatol. 2014 May-Jun;32(3):315-23. Epub 2014 Feb 11. PMID 24529163

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RA Subjects/ Infliximab 3 mg/kg
Started | 728
Completed | 597
Not Completed | 131
Not completed — Subject or treating physician's choice | 131

BASELINE CHARACTERISTICS:
Arm/Group | RA Subjects/ Infliximab 3 mg/kg
Number analyzed (Participants) | 728
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 571
  Male | 157
Time since diagnosis [Mean (Standard Deviation); unit: years] — Data available for 703 participants.
  years | 9.0 (8.99)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Raw Disease Activity Score for 28 Joint Swollen and Tender Joint Count (DAS28) by Age
Description: Results are reported as the mean DAS28 raw score at Baseline. DAS28 is a unit scale from 2.0 (best value) to 10.0 (worst value). The relationship between Baseline Raw DAS28 and Baseline age (see Baseline Characteristics) is reported in the statistical analysis.
Time Frame: At Baseline
Population: Efficacy evaluable population included all subjects who were enrolled and received at least one dose of study medication and with non-missing efficacy data at Baseline and at least one follow-up visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RA Subjects/ Infliximab 3 mg/kg
Number analyzed (Participants) | 662
Score on a scale | 5.2 (1.15)
Statistical Analysis 1: Comparison: RA Subjects/ Infliximab 3 mg/kg; Relationship between baseline DAS28 and age (prior to infliximab therapy); Test type: Superiority or Other; p = 0.0003, Test for non-zero correlation; Pearson Product Moment Correlation = 0.1402

2. Primary Outcome: Baseline Raw DAS28 by Time Since Diagnosis
Description: Results are reported as the mean DAS28 raw score at Baseline. DAS28 is a unit scale from 2.0 (best value) to 10.0 (worst value). The relationship between Baseline Raw DAS28 and time since diagnosis is reported in the statistical analysis.
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RA Subjects/ Infliximab 3 mg/kg
Number analyzed (Participants) | 662
Score on a scale | 5.2 (1.15)
Statistical Analysis 1: Comparison: RA Subjects/ Infliximab 3 mg/kg; Relationship between baseline DAS28 and time since diagnosis (prior to infliximab therapy); Test type: Superiority or Other; p = 0.7991, Test for non-zero correlation; Pearson Product Moment Correlation = -0.01

3. Primary Outcome: Baseline Raw DAS28 by Gender
Description: Results are reported as the mean DAS28 raw score at Baseline. DAS28 is a unit scale from 2.0 (best value) to 10.0 (worst value). The relationship between Baseline Raw DAS28 and Baseline gender (see Baseline Characteristics) is reported in the statistical analysis.
Time Frame: At Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | RA Subjects/ Infliximab 3 mg/kg | Male | Female
Number analyzed (Participants) | 662 | 140 | 522
Score on a scale | 5.2 (1.15) | 5.23 (1.11) | 5.19 (1.16)
Statistical Analysis 1: Comparison: Male vs Female; Relationship between baseline DAS28 and gender (prior to infliximab therapy); Test type: Superiority or Other; p = 0.7152, ANOVA; The association between Baseline DAS28 and gender is based on a one-way Anova

4. Primary Outcome: Baseline Raw DAS28 by Country of Residence
Description: Results are reported as the mean DAS28 raw score at Baseline. DAS28 is a unit scale from 2.0 (best value) to 10.0 (worst value). The relationship between Baseline Raw DAS28 and Baseline Characteristic is reported in the statistical analysis.
Time Frame: At Baseline
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Austria | Belgium | Denmark | France | Germany | Greece | Italy | Netherlands | Norway | Poland | Portugal | Sweden
Number analyzed (Participants) | 55 | 73 | 24 | 104 | 67 | 78 | 32 | 17 | 41 | 51 | 20 | 100
Score on a scale | 5.38 (0.90) | 5.43 (1.22) | 4.57 (1.16) | 4.97 (1.12) | 5.38 (1.23) | 5.15 (1.14) | 5.03 (1.05) | 5.07 (1.23) | 5.39 (1.13) | 5.83 (0.87) | 5.08 (1.48) | 4.96 (1.09)
Statistical Analysis 1: Comparison: Austria vs Belgium vs Denmark vs France vs Germany vs Greece vs Italy vs Netherlands vs Norway vs Poland vs Portugal vs Sweden; Relationship between baseline DAS28 and country of residence (prior to infliximab therapy); Test type: Superiority or Other; p < 0.0001, ANOVA; Relationship between DAS28 and Country of Residence was based on a 1-way ANOVA calculated as P-value

5. Primary Outcome: Baseline Raw DAS28 by Previous Anti-Tumor Necrosis Factor (Anti-TNF) Therapy
Description: Results are reported as the mean DAS28 raw score at Baseline. DAS28 is a unit scale from 2.0 (best value) to 10.0 (worst value). The relationship between DAS28 and baseline characteristic is reported in the statistical analysis.
Time Frame: At Baseline
Population: All efficacy evaluable subjects (n=662) included subjects with early RA not yet treated with anti-TNF (n=76), subjects with established RA not yet treated with anti-TNF (n=447), and subjects with RA who failed or did not tolerate another anti-TNF (n=123). Some subjects could not be classified into any subgroup due to missing diagnosis dates.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Early RA, Not Treated With Anti-TNF: Subjects with early RA not yet treated with an anti-TNF.
- Established RA, Not Treated With Anti-TNF: Subjects with established RA not yet treated with an anti-TNF.
- Established RA, Failed/Did Not Tolerate Another Anti-TNF: Subjects with established RA having failed or not tolerated another anti-TNF.
Arm/Group | RA Subjects/ Infliximab 3 mg/kg | Early RA, Not Treated With Anti-TNF | Established RA, Not Treated With Anti-TNF | Established RA, Failed/Did Not Tolerate Another Anti-TNF
Number analyzed (Participants) | 662 | 76 | 447 | 123
Score on a scale | 5.2 (1.15) | 5.3 (1.16) | 5.2 (1.14) | 5.3 (1.16)
Statistical Analysis 1: Comparison: RA Subjects/ Infliximab 3 mg/kg; Relationship between Baseline DAS28 and previous anti-TNF therapy (all subjects, prior to infliximab therapy); Test type: Superiority or Other; Mean Baseline DAS28 Raw Score = 5.2, 95% CI [5.1 to 5.3], Standard Deviation 1.15
Statistical Analysis 2: Comparison: Early RA, Not Treated With Anti-TNF; Relationship between Baseline DAS28 and previous anti-TNF therapy (subjects with early RA, not treated with anti-TNF; prior to infliximab therapy); Test type: Superiority or Other; Mean Baseline DAS28 Raw Score = 5.3, 95% CI [5.0 to 5.5], Standard Deviation 1.16
Statistical Analysis 3: Comparison: Established RA, Not Treated With Anti-TNF; Relationship between Baseline DAS28 and previous anti-TNF therapy (subjects with established RA not treated with anti-TNF; prior to infliximab therapy); Test type: Superiority or Other; Mean Baseline DAS28 Raw Score = 5.2, 95% CI [5.1 to 5.3], Standard Deviation 1.14
Statistical Analysis 4: Comparison: Established RA, Failed/Did Not Tolerate Another Anti-TNF; Relationship between Baseline DAS28 and previous anti-TNF therapy (subjects with established RA who failed or did not tolerate another anti-TNF; prior to infliximab therapy); Test type: Superiority or Other; Mean Baseline DAS28 Raw Score = 5.3, 95% CI [5.1 to 5.5], Standard Deviation 1.16

ADVERSE EVENTS:
Arm/Group | Infliximab 3 mg/kg
Serious Adverse Events (participants affected / at risk) | 40/721
Other Adverse Events (participants affected / at risk) | 0/721
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Infliximab 3 mg/kg (N=721)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
CHILLS (General disorders) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1)
HYPERTHERMIA (General disorders) | 1 (1)
INFUSION RELATED REACTION (General disorders) | 2 (4)
PYREXIA (General disorders) | 1 (1)
CHOLECYSTITIS (Hepatobiliary disorders) | 2 (2)
HYPERSENSITIVITY (Immune system disorders) | 1 (1)
BRONCHOPNEUMONIA (Infections and infestations) | 1 (1)
CELLULITIS (Infections and infestations) | 1 (1)
DISSEMINATED TUBERCULOSIS (Infections and infestations) | 1 (1)
ERYSIPELAS (Infections and infestations) | 1 (1)
INFECTION (Infections and infestations) | 1 (1)
MASTITIS (Infections and infestations) | 1 (1)
PNEUMOCYSTIS JIROVECI PNEUMONIA (Infections and infestations) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2)
PNEUMONIA LEGIONELLA (Infections and infestations) | 1 (1)
PYELONEPHRITIS (Infections and infestations) | 1 (1)
SALMONELLOSIS (Infections and infestations) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
DEVICE FAILURE (Injury, poisoning and procedural complications) | 1 (1)
SYNOVIAL RUPTURE (Injury, poisoning and procedural complications) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 1 (1)
INVESTIGATION (Investigations) | 1 (1)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OESOPHAGEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SPEECH DISORDER (Nervous system disorders) | 1 (1)
ALVEOLITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1 (1)
JOINT PROSTHESIS USER (Social circumstances) | 1 (1)
HERNIA REPAIR (Surgical and medical procedures) | 1 (1)
HYPERTENSION (Vascular disorders) | 1 (1)
PHLEBITIS (Vascular disorders) | 1 (1)
THROMBOSIS (Vascular disorders) | 2 (2)
VENOUS THROMBOSIS LIMB (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. If the parties disagree on the communication, the investigator and the sponsor's representative will meet for the purpose of making a good faith effort to discuss and resolve any such issues or disagreement.